CLINICAL TRIAL: NCT06725303
Title: Excimer Light Versus Blue Light in the Treatment of Inflammatory Acne, a Split Face Randomized Controlled Trial.
Brief Title: Excimer Light Versus Blue Light in Acne
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, University doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lights in acne treatment
Record Dates: First submitted 2024-12-08; First posted 2024-12-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Lasers, Excimer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Excimer light (Experimental): Light energy
  Interventions: Device: Excimer
- Blue light (Active Comparator): Light energy
  Interventions: Device: Excimer

INTERVENTIONS:
Device: Excimer — Light energy

SUMMARY:
The aim is to assess the efficacy and safety of Excimer Light versus blue light in the treatment of inflammatory acne.

DETAILED DESCRIPTION:
The use of new light energy in inflammatory acne

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate inflammatory acne lesions

Exclusion Criteria:

* Pregnancy during the first trimester

  * Female patients with a medical history of PCO
  * Topical and systemic treatment within the last month and systemic retinoids for 6 months
  * Patients on systemic steroid treatment or hormonal therapy
  * Severe systemic illness or malignancy
  * Photosensitivity
  * Scarring acne vulgaris

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of comedones, papules and pustules | 2 months
  number of lesions